CLINICAL TRIAL: NCT07045649
Title: Association Between Performance in the 1-Minute Sit-To-Stand Test and Clinical and Functional Outcomes of Patients Hospitalized for Heart Failure - Prospective Observational Study
Brief Title: Association Between the Sit-To-Stand Test and the Prognosis of Patients With Heart Failure
Status: Recruiting | Type: Observational
Sponsor: Centro Universitário Augusto Motta (Other)
Responsible Party: Sponsor
Other Study IDs: 87791825.8.0000.5235
Record Dates: First submitted 2025-05-12; First posted 2025-07-01 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Heart Failure; Heart Failure NYHA Class IV; Heart Failure; With Decompensation; Heart Failure NYHA Class III; Heart Failure NYHA Class II
Keywords: Functional Status; Hospitalization; Prognosis
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1-minute sit-to-stand test: The 1-minute sit-to-stand test will be assessed upon discharge from the Cardiac Intensive Care Unit. It may be assessed up to 48 hours after discharge from the unit. It will be performed on a standardized 46.0 cm chair without armrests, placed against the wall. Participants will be seated in the chair, without support, with their knees and hips at 90° flexion, with their feet parallel to the floor and their arms crossed over their chest. Participants will be instructed to stand up and sit down as quickly as possible without using their arms for 1 minute and will be instructed to stop whenever they wish. However, they must return as quickly as possible, since the goal is to complete as many repetitions as possible in 1 minute. Vital signs and dyspnea and leg fatigue will be assessed using the Modified Borg Scale before and after the test. A repetition will be identified as standing up completely straight and returning to the sitting position.
  Interventions: Diagnostic Test: 1-minute sit-to-stand test

INTERVENTIONS:
Diagnostic Test: 1-minute sit-to-stand test — The 1-minute sit-to-stand test will be assessed upon discharge from the Cardiac Intensive Care Unit. It may be assessed up to 48 hours after discharge from the unit. It will be performed on a standardized 46.0 cm chair without armrests, placed against the wall. Participants will be seated in the chair, without support, with their knees and hips at 90° flexion, with their feet parallel to the floor and their arms crossed over their chest. Participants will be instructed to stand up and sit down as quickly as possible without using their arms for 1 minute and will be instructed to stop whenever they wish. However, they must return as quickly as possible, since the goal is to complete as many repetitions as possible in 1 minute. Vital signs and dyspnea and leg fatigue will be assessed using the Modified Borg Scale before and after the test. A repetition will be identified as standing up completely straight and returning to the sitting position.

SUMMARY:
Introduction: Heart failure (HF), among cardiovascular diseases, is the disease that has been increasing its incidence and prevalence the most in recent years in the world population, due to the aging of the population. In addition, HF is the most frequent hospital diagnosis in the elderly, and is the main cause of hospitalization, with significant expenditure in public and private health care worldwide. Some functional tests have been used to predict the prognosis in patients with HF, however, the use of the 1-minute sit-to-stand test (SST1) to predict prognosis in HF has little scientific evidence, due to the lack of studies found in the literature for this population. Thus, the present study aims to evaluate the association between SST1 at discharge from the Cardio Intensive Care Unit (ICU) and the clinical outcome after 90 days in patients hospitalized for decompensated heart failure (DHF). Methods: This is a prospective cohort study analyzing the association between performance on the TSL1 and clinical outcome in patients hospitalized for DHF from June 2025 to October 2025. Sociodemographic, family, social, and clinical data will be collected from the participants, after which the TSL1 will be performed. The outcome of death and hospital readmission within 90 days after discharge from the ICU will be identified through telephone contact, which will be carried out by the researcher. Expected results: It is expected that from the results of this study it will be possible to understand whether performance on the TSL1 predicts clinical outcome for patients hospitalized for DHF and that it will even be possible to determine a cutoff point capable of predicting the outcomes of interest.

DETAILED DESCRIPTION:
This is a prospective cohort study analyzing the association between TSL1 performance and clinical and functional outcomes within 90 days after discharge of patients who were hospitalized for CDI between June 2025 and October 2025. Data will be collected by the researcher and the institution's senior physiotherapist team, and the team will be trained to reduce the risk of bias. A document form will be made available for completion during the evaluation, and sociodemographic data will also be collected from the electronic medical record.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with CDI;
* Over 18 years of age;
* With an Intensive Care Unit Mobility Scale (IMS) > 4 at discharge from the ICU;
* Able to sit and stand up from a chair without support from the upper limbs (ULs) will be included in the study.

Exclusion Criteria:

* Patients with cognitive alterations;
* Level of consciousness, with [RASS (Richmond Agitation and Sedation Scale) >+1 or <-2 and Glasgow <13 (Coma Scale)], neurological and orthopedic, which compromise the understanding and performance of the assessment will be excluded;
* Patients with advanced invasive ventilatory and circulatory support or in cardiogenic shock.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with CDI
Sampling Method: Non-Probability Sample
Enrollment: 68 (Estimated)
Dates: Start 2025-07-16 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Occurrence of mortality for any cause within 90 days after discharge from the Cardiac Intensive Care Unit (ICU) in patients hospitalized for decompensated heart failure (DHF). | 90 days after discharge from the ICU
Number of readmission for any cause within 90 days after discharge from the Cardiac Intensive Care Unit (ICU) in patients hospitalized for decompensated heart failure (DHF). | 90 days after discharge from the ICU

SECONDARY OUTCOMES:
All-cause mortality within 90 days of discharge | 90 days after discharge from the ICU
Readmission due to HF within 90 days after discharge | 90 days after discharge from the ICU
Total number of days alive outside the hospital (days alive after discharge by time from occurrence to event) in the first 90 days after discharge | 90 days after discharge from the ICU
Functional performance at the time of discharge from the ICU according to the IMS - Intensive Care Unit Mobility Scale | In the 48 hours prior to discharge from the ICU
Correlation between TSL-1 performance and other functional markers at discharge (FSS-ICU, IMS and handgrip strength) | In the 48 hours prior to discharge from the ICU

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitário Pedro Ernesto, Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No